CLINICAL TRIAL: NCT03351283
Title: Effect of Moderate vs Severe Sodium Restriction on Brain Natriuretic Peptide in Patients With Heart Failure and Reduced Ejection Fraction
Brief Title: Effect of Sodium Intake on Brain Natriuretic Peptide Levels in Patients With Heart Failure
Acronym: SODA-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Eduardo Almeida Gutiérrez, Dr, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sodium and BNP
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Diet, Sodium-Restricted; Heart Failure, Systolic; Natriuretic Peptide, Brain; Clinical Trial
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe sodium restriction (Experimental): Patients will be assigned to a diet with two grams of sodium. The nutritionist will be responsible for calculating diets appropriate to the needs of each patient. The diet will not have the intention to modify the weight of the patient but only to indicate the menus that the patients will follow. All the patients will be explained the diet. Patients will be allowed a maximum intake of 1.5 liters of water per day, including the liquid of soups, juices and drinks; This will be explained in detail to the patients.
  The diets will be identical in calories according to the weight of the patient. The only difference in diets will be the sodium content, which will be 2 grams of sodium vs. 3 grams of sodium.
  Interventions: Other: Severe sodium restriction
- Moderate sodium restriction. (Active Comparator): Patients will be assigned to a diet with three grams of sodium.
  Interventions: Other: Moderate sodium restriction

INTERVENTIONS:
Other: Severe sodium restriction — Patients will be assigned to a diet with sodium restriction of two grams.
  Arms: Severe sodium restriction
Other: Moderate sodium restriction — Patients will be assigned to a diet with sodium restriction of three grams.
  Arms: Moderate sodium restriction.

SUMMARY:
The SODA-HF trial is a randomized, double-blind, controlled trial to evaluate the effect of moderate to severe sodium restriction on brain natriuretic peptide in patients with heart failure and reduced ejection fraction (less than 40%).

Secondary outcomes are quality of life, NYHA functional class, glomerular filtration rate, renin plasmatic activity, aldosterone and composite clinical outcome (all-cause mortality and cardiovascular hospitalization)

DETAILED DESCRIPTION:
Allocation: Those patients who meet the selection criteria will go to the nutritionist who will make the assignment to one of the sodium restriction groups.

Generation of the sequence: patients will be assigned to the two groups based on a table of random numbers generated by a statistical analysis program. Blocks of 10 will be used.

Mechanism of concealment of the assignment: the nutritionist will be the only person who will know to which group the patient was assigned, the patient will not know to which group was assigned, neither will the researcher know. The person in charge of measuring the results will also be blinded.

Description of the intervention: the nutritionist will be the one to calculate diets appropriate to the needs of each of the patients. Patients will be allowed a maximum intake of 1.5 liters of water per day, including the liquid of soups, juices and drinks; This will be explained in detail to the patients. The diets will be identical in calories according to the weight of the patient. The only difference in diets will be the sodium content, which will be 3 grams of sodium vs. 2 grams of sodium.

Blinding: The patients, the researcher and those responsible for measuring the results will be blinded to the assignment of the intervention. Patients will not know which group they have been assigned to since they will not know the sodium content of the diet nor will they be aware of what diet the other patients were assigned to. Those responsible for conducting laboratory studies will not know to which group the patients have been assigned.

Blinding may be opened in the event that a patient suffers a severe adverse effect.

Follow-up: After assignment of the intervention, the patients will be cited at 6, 12 and 20 weeks. In Nutriology visits, the adherence of the intervention will be evaluated by means of a 24-hour diet reminder. According to the results obtained, the nutritionist will make recommendations in the diet to maintain a sodium intake of 3000 or 2000 mg according to the group to which hte patient has been assigned.

At the end of the intervention the natriuretic peptide value will be determined, as well as plasma activity of renin, aldosterone, GFR and the composite clinical outcome (all-cause mortality and cardiovascular hospitalization).

If a patient is hospitalized during the study, he will follow the treatment indicated by his treating doctor. Once the patient is discharged from the hospital, he will continue with previously scheduled follow-up appointments. If the sampling scheduled during the study coincides with an episode of unplanned hospitalization, the patient will wait until the patient has completed at least 4 weeks after discharge to take the corresponding samples.

If any patient dies during the study, he will be eliminated from the primary objective which is the determination of natriuretic peptide.

Monitoring of the study. Monitoring of information: Given that the study will be conducted in a single center, it is considered that a data monitoring committee will not be necessary.

Monitoring of patient safety: During the scheduled medical visits, a complete physical examination will be carried out with detailed attention to the signs and symptoms of heart failure. Weight, height, heart rate and systemic blood pressure will be measured. If a patient presents symptoms of heart failure exacerbation, he will be taken to the emergency department for a complete evaluation and adjustment of treatment.

According to the Mexican Official Norm 012-SSA3-2012, it will be considered adverse effect to the set of signs and symptoms not calculated and unexpected that appear in a research subject, and that potentially represent a risk to his health. If an adverse effect occurs, it will be notified no later than the business day following the corresponding Research Committee. In case of a severe adverse event (one that endangers the patient's life), the corresponding Research Committee will be notified immediately.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of stable heart failure and decreased left ventricular ejection fraction. Such definition will contemplate the following:

1. Patients should have an echocardiogram of maximum 6 months old with a left ventricular ejection fraction of less than 40%.
2. Functional class I, II or III of the NYHA
3. Optimal medical treatment which should include: an angiotensin converting enzyme inhibitor or angiotensin receptor blocker ARA, and a beta-blocker; or inability to tolerate these medications.
4. No changes in pharmacological treatment in the last 4 weeks.
5. Systolic blood pressure greater than or equal to 90 mmHg.
6. Informed consent to participate in the study.

Exclusion Criteria:

A hospitalization for heart failure less than one month ago. Chronic kidney disease: glomerular filtration rate estimated by the formula of CKD-EPI <30 ml / min / 1.73 m2.

Hyponatremia: Sodium less than 130 mmol / l. Anemia: Hemoglobin less than 10 g / dl. Patients who will be taken to any type of intervention in the next 12 months in order to improve ventricular function, such as percutaneous coronary intervention or surgical revascularization Any valvulopathy of severe degree. Dementia Cancer Patients who have planned change of address in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Brain natriuretic peptide | 20 weeks
  Brain natriuretic peptide (NT-proBNP) will be compared at the end of the intervention.

SECONDARY OUTCOMES:
Improvement in Quality of life | 20 weeks
  Quality of life will be compared with the Minnesota Living with Heart Failure Questionnaire. This is a self-applied questionnaire that contains 21 items, a total score and two dimensions: physical and emotional. The response options range from 0, which indicates unaffected quality of life, to 5, which indicates the maximum impact on the quality of life. The range of values of the questionnaire in general is 0-105; the physical dimension is 0-40; The emotional dimension is 0-25. In this study we will compare the overall result and the two dimensions.
Measured glomerular filtration rate | 20 weeks
  Measured glomerular filtration rate will be assessed with 24-hour creatinine clearance.
Renin plasmatic activity | 20 weeks
  Renin plasmatic activity will be assessed with ELISA.
Aldosterone | 20 weeks
  Aldosterone will be assessed with ELISA.
Composite clinical outcome | 20 weeks
  All-cause mortality or cardiovascular hospitalizations
NYHA functional class | 20 weeks
  The range of the NYHA functional class is I to IV, where I is the patient with the best functional class and IV is a patient with the worst functional class.

OTHER OUTCOMES:
Estimated glomerular filtration rate | 20 weeks
  Glomerular filtration rate will be assessed with the CKD-EPI equation.

CONTACTS AND LOCATIONS:
Overall Officials: Juan B Ivey-Miranda, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de Cardiología, Centro Médico Nacional Siglo XXI, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
IPD will not be freely available but can be shared to certain investigators.

REFERENCES:
- [Derived] Ivey-Miranda JB, Almeida-Gutierrez E, Herrera-Saucedo R, Posada-Martinez EL, Chavez-Mendoza A, Mendoza-Zavala GH, Cigarroa-Lopez JA, Magana-Serrano JA, Rivera-Leanos R, Trevino-Mejia A, Revilla-Matute C, Flores-Umanzor EJ, Espinola-Zavaleta N, Orea-Tejeda A, Garduno-Espinosa J, Saturno-Chiu G, Rao VS, Testani JM, Borrayo-Sanchez G. Sodium restriction in patients with chronic heart failure and reduced ejection fraction: A randomized controlled trial. Cardiol J. 2023;30(3):411-421. doi: 10.5603/CJ.a2021.0098. Epub 2021 Sep 7. PMID 34490604